CLINICAL TRIAL: NCT02918916
Title: Effect of Phototherapy Applied During Combined Training on Performance and Post-exercise Recovery: Study Protocol of a Randomized Controlled Trial by Stratified Sample, Double-blind, Placebo-controlled
Brief Title: Phototherapy Applied During Combined Training
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: São Paulo State University (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2015/25219-0
Record Dates: First submitted 2016-09-26; First posted 2016-09-29 (Estimated); Last update posted 2016-09-29 (Estimated); Status verified 2016-09

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Phototherapy; Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Active phototherapy group (Experimental): Phototherapy will be applied between sprint and squat training (exactly 10 minutes before squat training).
  Active phototherapy will be applied by a trained therapist using a MR4 LaserShower 50 4D emitter (Multi Radiance Medical, USA), bilaterally to six sites of the quadriceps (two centrally - rectus femoris and vastus intermedius; two laterally - vastus lateralis; two medially - vastus medially) in direct contact with the skin.
  The optical power will be calibrated before irradiation in each participant using a Thorlabs thermal power meter (Model S322C, Thorlabs, Newton, New Jersey, USA).
  Interventions: Other: Phototherapy
- Placebo phototherapy group (Placebo Comparator): Placebo will be applied between sprint and squat training (exactly 10 minutes before squat training). Placebo phototherapy will be applied by a trained therapist using a MR4 LaserShower 50 4D emitter (Multi Radiance Medical, USA), bilaterally to six sites of the quadriceps (two centrally - rectus femoris and vastus intermedius; two laterally - vastus lateralis; two medially - vastus medially) in direct contact with the skin. To receive active or placebo phototherapy the participant will be placed in the supine position.
  The same procedures as in the active phototherapy group will be applied to the placebo phototherapy group; however the emitter will be disabled.
  Interventions: Other: Placebo
- Control group (No Intervention): Passive recovery will be applied between sprint and squat training (exactly 10 minutes before squat training). During the period when the other groups are receiving recovery strategies, the control group participants will remain seated for passive recovery, supervised by an independent therapist.

INTERVENTIONS:
Other: Phototherapy — The dosage applied will be 30 Joules per site (180 Joules per muscle). Parameters are described in the attached document.
  Other Names: Low-level laser therapy; Light-emitting diode
  Arms: Active phototherapy group
Other: Placebo — The same procedures as in the active phototherapy group will be applied to the placebo phototherapy group; however the emitter will be disabled.
  Arms: Placebo phototherapy group

SUMMARY:
Introduction: Recent studies have shown positive results from the application of phototherapy for the improvement of performance and acceleration of the recovery process both in the application before and after exercise. However, the effects of phototherapy during combined training and after a primary adaptation process remain unclear.

Research objectives: The primary objective of the study is to analyze and compare the effects of phototherapy using different light sources (laser and light emmiting diode - LED) interacting with combined training on clinical, functional, and psychological outcomes and vascular endothelial growth factor. The secondary objective is to compare the benefits provided by phototherapy in participants with different levels of training adaptation.

Design: A controlled trial, double-blind, placebo-controlled will be conducted with stratified randomization and concealed allocation.

Participants and Setting: After fulfilling the eligibility criteria, forty-five male participants will participate in the study.

Procedure: In phase 1, the participants will perform six-weeks of combined training (sprints and squats). In phase 2, participants will be allocated, through stratified randomization (based on adaptation capacity to training), into three groups: active phototherapy group (AG), placebo phototherapy group (PG), and control group (CG). A new six-week training period will then start. In this phase the participants will carry out training normally with the adjusted loads and between sprints and squats will receive the recovery strategy related to the group to which they belong.

Intervention: Active and placebo phototherapy will be applied by a trained therapist, between sprints and squats. During the period of recovery strategies for the AG and PG, the CG participants will remain seated for passive recovery, supervised by an independent therapist.

Measurements: The measurements include clinical, functional, and psychological outcomes and vascular endothelial growth factor.

DETAILED DESCRIPTION:
Introduction: Recent studies have shown positive results from the application of phototherapy for the improvement of performance and acceleration of the recovery process both in the application before and after exercise. However, the effects of phototherapy during combined training and after a primary adaptation process remain unclear.

Research objectives: The primary objective of the study is to analyze and compare the effects of phototherapy using different light sources (laser and LEDs) interacting with combined training on clinical, functional, and psychological outcomes and vascular endothelial growth factor. The secondary objective is to compare the benefits provided by phototherapy in participants with different levels of training adaptation.

Design: A controlled trial, double-blind, placebo-controlled will be conducted with stratified randomization and concealed allocation.

Participants and Setting: After fulfilling the eligibility criteria, forty-five male participants will participate in the study. The inclusion criteria include: healthy male, aged between 18-30 years who agree to participate in the study. Participants with the following will be excluded from the study: presence of anemia, inflammation, diabetes, history of metastasis or muscle injury in the lower limbs or spine in the previous six months, and occurrence of musculoskeletal injury during the study.

Procedure: In phase 1, the participants will perform six-weeks of combined training (sprints and squats). In phase 2, participants will be allocated, through stratified randomization (based on adaptation capacity to training), into three groups: active phototherapy group (AG), placebo phototherapy group (PG), and control group (CG). A new six-week training period will then start. In this phase the participants will carry out training normally with the adjusted loads and between sprints and squats will receive the recovery strategy related to the group to which they belong.

Intervention: Active and placebo phototherapy will be applied by a trained therapist, between sprints and squats, bilaterally to six sites of the quadriceps in direct contact with the skin. The dosage applied will be 30J per site. The same procedures as the AG will be applied to the PG, however the emitter will be disabled. During the period of recovery strategies for the AG and PG, the CG participants will remain seated for passive recovery, supervised by an independent therapist.

Measurements: The measurements include clinical (muscle soreness, pain threshold, perception of exertion, and perception of recovery), functional (squat strength and power, maximal voluntary isometric contraction, maximal incremental test, squat jump, and sprint test), and psychological (self-assessments of readiness for exercise, fatigue, vigor, pain, and belief of intervention effectiveness) outcomes and vascular endothelial growth factor.

Analysis: For analysis of functional outcomes, data normality will be checked by the Kolmogorov-Smirnov test with changes from baseline followed by the Student T test for comparisons. For other outcomes, sphericity of the data will be tested by the Mauchly's test. In case of violation of the sphericity assumption, Greenhouse-Geisser corrections will be used. Data will be analyzed using repeated-measures analysis of variance (Bonferroni's test will be performed when required), which provide information on time, group, and interaction effects. A significance level of 5% will be assumed for all statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Healthy (self-report);
* Male gender;
* Aged between 18-30 years;
* Agreement to participate through signed statement of informed consent

Exclusion Criteria:

* Presence of anemia, inflammation, or diabetes;
* History of metastasis.
* History of muscle injury in the lower limbs or spine in the previous six months;
* Occurrence of musculoskeletal injury during the study.

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2017-01; Primary Completion 2018-03 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Change from 6-week Maximal voluntary isometric contraction at 12-week of training | Change between 6-week and 12-week of training
  Prior to the MVIC evaluation, participants will conduct a warm up consisting of 10 repetitions of knee flexion-extension at 180°.s-1 throughout the range of motion. The MIVC will be determined by the highest maximal isometric torque over three contractions of five seconds at 60° of knee flexion (with 0° corresponding to the maximum extension). The repetitions will be separated by a 2-minute rest interval. Participants will be instructed to perform maximal contractions and verbally encouraged by the researcher during the evaluation.

SECONDARY OUTCOMES:
Strength and power test | Baseline, after 6-week, after 13-week of training
  Strength and power tests will be carried out in vertical squat equipment with a guided bar.
Maximum oxygen consumption (VO2max) | Baseline, after 6-week, after 13-week of training
  The maximum oxygen consumption (VO2max) will be determined on a treadmill using an incremental protocol.
  Gas analysis will be measured continuously and the average value of every 30 seconds recorded (VO2000, MedGraphics, Minnesota, USA).
Squat jump | Baseline, after 6-week, after 13-week of training
  To perform the squat jump test, the participant will remain with the sole of their feet in contact with the jump platform (Multisprint, Hidrofit, Brazil), legs at 90° of flexion, hands on hips, trunk upright and without previous movements. The participant will perform a jump keeping their legs straight (180°) and touch the platform again.
  Each participant will perform three complete tests with a rest interval of 30 seconds between each repetition. The best measure of the tests will be adopted.
Sprint test | Baseline, after 6-week, after 13-week of training
  To perform the sprint test, participants will perform three maximum sprints exceeding 30 meters with rest intervals of 3-minutes. Performance times at 10, 20 and 30 meters will be recorded by photocells (Multisprint, Hidrofit, Brazil). The average of the two best tests will be adopted. Participants will be encouraged verbally during the test.
Muscle soreness | Baseline, 5-week, after 6-week, 12-week, after 13-week of training
  Values of muscle soreness will be obtained through a visual analog scale (VAS), with 10-points, with 'zero' corresponding to absence of soreness and '10' to the maximum level supported by the participant, as described previously. Participants will be asked about the presence of soreness in the lower limbs.
Pain threshold | Baseline, 5-week, after 6-week, 12-week, after 13-week of training
  To assess the pain threshold, pressure algometry will be applied at five specific sites of the quadriceps. The participant will be placed in the supine position and the markers will be carried out in the dominant leg. The sites will be located using the reference system, which primarily identifies two anatomic points: anterior superior iliac spine (ASIS) and upper pole of the patella (UPP). Thus, the sites assessed will be: 15 cm distal to the ASIS, 4 cm proximal to the UPP, mean point between the ASIS and UPP, and 2 cm lateral and medial to the mean point.
  Pain threshold will be defined in Kgf through the minimal pressure required to induce a pain sensation or discomfort. Participants will be instructed to signal when the pressure sensation becomes discomfort. The pressure will not exceed 2.55 Kgf.
Perception of exertion | 5-week, 12-week of training
  The level of exertion reported by participants will be assessed using the Borg Scale (6-20 points), with 'six' corresponding to 'very easy' and '20' to 'exhaustive'. Participants will be asked about their perception of exertion in the upper and lower limbs.
Perception of recovery | 5-week, 12-week of training
  Perception of recovery will be assessed by a 10-point Likert Scale, with 'one' corresponding to 'not recovered' and '10' to 'fully recovery'.
Psychological questionnaire | Baseline, before 5-week, before 12-week of training
  Participants will complete a psychological questionnaire that aims to document, subjectively, the readiness for exercise, fatigue, vigor, sleepiness, and pain. Participants will be instructed to mark an "X" on a 10-cm visual analog scale between two extremes, with 'zero' corresponding to 'least possible' and '10' 'most possible' for each rating.
Belief questionnaire | After 6-week, after 13-week of training
  After phase 1, participants will answer a belief questionnaire to measure their 'belief' in the effectiveness of the technique. Participants will be instructed to mark an "X" on a 5-point Likert Scale, with 'zero' corresponding to 'not effective' and 'ten' to 'extremely effective'.
  After application of the recovery techniques, the participants will complete a similar questionnaire to measure their perceived effectiveness of the technique.
Vascular endothelial growth factor | Baseline, after 6-week, after 13-week
  To analyze the vascular endothelial growth factor (VEGF) 10 ml of blood will be collected. Plasma from this sample will be stored at -80°C for later analysis. The plasma level of VEGF will be analyzed using the ELISA method in duplicate (enzyme-linked immunosorbent assays) following the manufacturer's instructions (RayBio, Norcross, GA, USA).

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Pastre, PhD, Principal Investigator — Univ Estadual Paulista

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- Available data/document: Tables. Training program, Phototherapy parameters, Time point of outcomes — https://pt.scribd.com/document/325401697/Documents-ClinicalTrials-ID-2015-25219-0